CLINICAL TRIAL: NCT03414840
Title: Assessment of Change in Atherosclerotic Plaque by Serial CCTA
Acronym: ACROSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Collaborators: Chong Kun Dang Pharmaceutical Corp. (Industry)
Responsible Party: Principal Investigator, Hyuk-Jae Chang, Professor, Yonsei University
Other Study IDs: 2017-2669-001
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Coronary Arteriosclerosis
Keywords: coronary artery disease; coronary computed tomography angiography; statins; coronary atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atorvastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Atorvastatin — Patients diagnosed with coronary artery disease by CCTA be enrolled. Among enrolled patients, patients who is indicated to statin treatment according to the current ACC/AHA guideline will be treated with atorvastatin.

SUMMARY:
Assessment of Change in AtheROSclerotic Plaque by Serial CCTA (ACROSS) is designed as a prospective observational study which aim is to demonstrate the effect of statins on coronary atherosclerosis, assessed by quantitative analysis of CCTA.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent clinically indicated CCTA (index CCTA)
* Mild to moderate stenosis (25-69%) on CCTA
* ≥1 clinical risk factors (Smoking, HTN, HDL<40, Premature FHx, M ≥45, F ≥55) for CAD

Exclusion Criteria:

* Acute coronary syndrome (unstable angina or MI)
* Positive (not equivocal) stress test
* Contraindications to statin

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent clinically indicated CCTA and confirmed to have coronary atherosclerosis will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Difference in percent change of total atheroma volume assessed by CCTA between statin-taking and statin-naïve group | 24 months
  Patients indicated with statin therapy according to current guideline will receive atorvastatin.

SECONDARY OUTCOMES:
Change of total atheroma volume at 24 months compared with baseline total atheroma volume | 24 months
  total atheroma volume assessed by CCTA

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk-Jae Chang, MD, PhD, Principal Investigator — Yonsei University
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No